CLINICAL TRIAL: NCT01949545
Title: An Open-Label, Single Arm, Phase 1 Study of the Pharmacokinetics and Safety of Carfilzomib in Subjects With Advanced Malignancies and Varying Degrees of Hepatic Impairment
Brief Title: Study of the Pharmacokinetics and Safety of Carfilzomib in Patients With Advanced Malignancies and Hepatic Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CFZ002; 20130402 (Other: Amgen)
Record Dates: First submitted 2013-09-06; First posted 2013-09-24 (Estimated); Results first posted 2016-10-21 (Estimated); Last update posted 2017-05-02 (Actual); Status verified 2017-04

CONDITIONS: Solid Tumors; Hematologic Malignancies; Hepatic Impairment
MeSH Terms: conditions — Hematologic Neoplasms | interventions — carfilzomib; WW Domain-Containing Oxidoreductase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Normal Hepatic Function (Experimental): Participants with normal hepatic function (bilirubin and aspartate aminotransferase (AST) ≤ the upper limit of normal (ULN)) received carfilzomib 20 mg/m² administered by intravenous (IV) infusion on days 1 and 2 of cycle 1, followed by a planned step-up to 27 mg/m² IV on days 8, 9, 15, and 16 of cycle 1. Participants who adequately tolerated dosing at 27 mg/m² in cycle 1 received carfilzomib 56 mg/m² IV on days 1, 2, 8, 9, 15, and 16 of cycle 2 and subsequent 28-day cycles until confirmed progressive disease (PD), unacceptable toxicity, withdrawal of consent, study closure, or death.
  Interventions: Drug: Carfilzomib
- Mild Hepatic Impairment (Experimental): Participants with mild hepatic impairment (bilirubin > 1-1.5 x ULN or AST > ULN, but bilirubin ≤ ULN) received carfilzomib 20 mg/m² administered by intravenous (IV) infusion on days 1 and 2 of cycle 1, followed by a planned step-up to 27 mg/m² IV on days 8, 9, 15, and 16 of cycle 1. Participants who adequately tolerated dosing at 27 mg/m² in cycle 1 received carfilzomib 56 mg/m² IV on days 1, 2, 8, 9, 15, and 16 of cycle 2 and subsequent 28-day cycles until confirmed progressive disease (PD), unacceptable toxicity, withdrawal of consent, study closure, or death.
  Interventions: Drug: Carfilzomib
- Moderate Hepatic Impairment (Experimental): Participants with moderate hepatic impairment (bilirubin > 1.5-3 x ULN, any AST) received carfilzomib 20 mg/m² administered by intravenous (IV) infusion on days 1 and 2 of cycle 1, followed by a planned step-up to 27 mg/m² IV on days 8, 9, 15, and 16 of cycle 1. Participants who adequately tolerated dosing at 27 mg/m² in cycle 1 received carfilzomib 56 mg/m² IV on days 1, 2, 8, 9, 15, and 16 of cycle 2 and subsequent 28-day cycles until confirmed progressive disease (PD), unacceptable toxicity, withdrawal of consent, study closure, or death.
  Interventions: Drug: Carfilzomib
- Severe Hepatic Impairment (Experimental): (Bilirubin > 3 × ULN; any AST) Participants with severe hepatic impairment (bilirubin > 3 x ULN; any AST) received carfilzomib 20 mg/m² administered by intravenous (IV) infusion on days 1 and 2 of cycle 1, followed by a planned step-up to 27 mg/m² IV on days 8, 9, 15, and 16 of cycle 1. Participants who adequately tolerated dosing at 27 mg/m² in cycle 1 received carfilzomib 56 mg/m² IV on days 1, 2, 8, 9, 15, and 16 of cycle 2 and subsequent 28-day cycles until confirmed progressive disease (PD), unacceptable toxicity, withdrawal of consent, study closure, or death.
  Interventions: Drug: Carfilzomib

INTERVENTIONS:
Drug: Carfilzomib — Carfilzomib was administered by IV injection over 30 minutes
  Other Names: Kyprolis® (carfilzomib) for Injection

SUMMARY:
The purpose of this study is to compare the safety and efficacy of carfilzomib, including measuring the amount of the study drug in the blood at certain times following dosing. This study is being done in people with varying degrees of liver function to see if they respond differently to the study drug.

ELIGIBILITY:
Key Inclusion Criteria:

1. Relapsed or progressive advanced malignancies (solid tumors or hematologic malignancies)
2. At least ≥ 2 prior treatment regimens for the underlying malignancy
3. Confirmed advanced solid tumor or hematologic malignancy
4. Measurable or evaluable disease
5. Clinical diagnosis of chronic hepatic impairment that is stable with no acute worsening of liver failure within one month prior to enrollment. Hepatic impairment will be assessed as per National Cancer Institute Organ Dysfunction Working Group Criteria (NCI-ODWG) schema and will fall into one of the following three categories:

   * Cohort 2 (mild): Bilirubin > 1-1.5 × upper limit of the normal range (ULN) or aspartate aminotransferase (AST) > ULN, but bilirubin ≤ ULN
   * Cohort 3 (moderate): ≥ 1.6-3 × ULN; any AST
   * Cohort 4 (severe): Bilirubin > 3 × ULN; any AST

   Exception to Inclusion Criterion #5 for Subjects with Normal Hepatic Function:

   All subjects enrolled with normal hepatic function (N=10) must meet all inclusion criteria as outlined with the exception of Inclusion Criterion

   #5, which should be substituted with the following criterion to be enrolled into the study:

   - Cohort 1 (normal hepatic function): Bilirubin ≤ ULN; AST ≤ ULN
6. Eastern Cooperative Oncology Group (ECOG) Performance Status 0-2
7. Left ventricular ejection fraction (LVEF) ≥ 40%
8. Adequate renal function (calculated creatinine clearance ≥ 30 mL/min)
9. Active congestive heart failure (New York Heart Association [NYHA] Class III to IV), symptomatic ischemia, conduction abnormalities uncontrolled by conventional intervention or myocardial infarction within the protocol-specified period prior to enrollment

Key Exclusion Criteria:

1. Subjects with symptomatic brain metastasis or central nervous system (CNS) disease
2. Significant neurotoxicity (Grade 2 with pain or higher) at the time of enrolment
3. Known human immunodeficiency virus (HIV), hepatitis B virus (HBV) and hepatitis C virus (HCV) infection (Exception: Subjects with chronic or cleared HBV and HCV infection and stable liver function tests [bilirubin, AST] will be allowed)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2013-10; Primary Completion 2015-08 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (11):
- United States (5):
  - Karmanos Cancer Institute, Detroit, Michigan
  - Duke Cancer Institute, Durham, North Carolina
  - Gabrail Cancer Center, Canton, Ohio
  - Tennessee Oncology, PLLC, Nashville, Tennessee
  - Evergreen Hematology and Oncology, Spokane, Washington
- Institut Gustave Roussy, Paris, Villejuif Cedex, France
- University Medical Centre Utrecht, Utrecht, Netherlands
- United Kingdom (4):
  - Northern Ireland Cancer Trials Centre - Queen's University Belfast TriaIs Centre, Belfast, Northern Ireland
  - Beatson West of Scotland Cancer Centre, Glasgow, Scotland
  - Velindre Hospital, Cardlff, Wales
  - Sir Bobby Robson Cancer Trials Research Centre, Newcastle

REFERENCES:
- [Derived] Brown J, Plummer R, Bauer TM, Anthony S, Sarantopoulos J, De Vos F, White M, Schupp M, Ou Y, Vaishampayan U. Pharmacokinetics of carfilzomib in patients with advanced malignancies and varying degrees of hepatic impairment: an open-label, single-arm, phase 1 study. Exp Hematol Oncol. 2017 Oct 3;6:27. doi: 10.1186/s40164-017-0086-1. eCollection 2017. PMID 29026685

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were assigned to 1 of 4 cohorts with varying degrees of hepatic impairment defined by the National Cancer Institute Organ Dysfunction Working Group Criteria (NCI-ODWG) schema for hepatic function.
  Completed indicates participants who completed the safety follow-up visit 30 days after the last dose of carfilzomib.
Groups:
- Severe Hepatic Impairment: Participants with severe hepatic impairment (bilirubin > 3 x ULN; any AST) received carfilzomib 20 mg/m² administered by intravenous (IV) infusion on days 1 and 2 of cycle 1, followed by a planned step-up to 27 mg/m² IV on days 8, 9, 15, and 16 of cycle 1. Participants who adequately tolerated dosing at 27 mg/m² in cycle 1 received carfilzomib 56 mg/m² IV on days 1, 2, 8, 9, 15, and 16 of cycle 2 and subsequent 28-day cycles until confirmed progressive disease (PD), unacceptable toxicity, withdrawal of consent, study closure, or death.
Period: Overall Study
Arm/Group | Normal Hepatic Function | Mild Hepatic Impairment | Moderate Hepatic Impairment | Severe Hepatic Impairment
Started | 11 | 17 | 14 | 4
Completed | 11 | 17 | 14 | 4
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Normal Hepatic Function | Mild Hepatic Impairment | Moderate Hepatic Impairment | Severe Hepatic Impairment | Total
Number analyzed (Participants) | 11 | 17 | 14 | 4 | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.5 (8.2) | 59.5 (9.1) | 61.0 (7.9) | 56.3 (10.9) | 61.8 (9.3)
Age, Customized [Number; unit: participants]
  < 65 years | 3 | 12 | 8 | 3 | 26
  ≥ 65 years | 8 | 5 | 6 | 1 | 20
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 8 | 5 | 3 | 18
  Male | 9 | 9 | 9 | 1 | 28
Race/Ethnicity, Customized [Number; unit: participants]
  Black | 0 | 1 | 1 | 0 | 2
  White | 11 | 13 | 13 | 4 | 41
  Not reported | 0 | 3 | 0 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration Time Curve From Time Zero to Last Concentration Measured (AUC0-last) of Carfilzomib 27 mg/m²
Description: The area under the curve from time zero (defined as the start of carfilzomib infusion) to the last concentration measured (AUC0-last) following intravenous administration of carfilzomib 27 mg/m² on day 16 of cycle 1 was calculated using a non-compartmental approach, from the individual plasma concentration profiles of carfilzomib.
Time Frame: Cycle 1 day 16, pre-dose, 15 minutes after the start of infusion, immediately (within 2 minutes) before the end of infusion, and at 5, 15, and 30 minutes and 1, 2, and 4 hours after the end of the infusion.
Population: Pharmacokinetic-evaluable population, defined as participants who received the intended carfilzomib dose (27 or 56 mg/m²) and who had plasma concentration versus time data for the estimation of each pharmacokinetic (PK) parameter by a non-compartmental analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Normal Hepatic Function | Mild Hepatic Impairment | Moderate Hepatic Impairment | Severe Hepatic Impairment
Number analyzed (Participants) | 10 | 14 | 9 | 0
ng*hr/mL | 378 (40.8) | 546 (39.2) | 477 (33.1) |
Statistical Analysis 1: Comparison: Normal Hepatic Function vs Mild Hepatic Impairment; To assess the effect of hepatic impairment relative to participants with normal hepatic function on AUC0-last an analysis of variance (ANOVA) of the log-transformed plasma PK parameters was performed. The ANOVA model included hepatic impairment as a fixed effect; Test type: Superiority or Other; p = 0.02232, ANOVA; Geometric Mean Ratio = 144.43, 95% CI 2-sided [111.48 to 187.12] — The geometric mean ratio was calculated by exponentiation of the differences in the least squares means, using log-transformed data, between the hepatic impairment cohort (test) and participants with normal hepatic function (reference)
Statistical Analysis 2: Comparison: Normal Hepatic Function vs Moderate Hepatic Impairment; To assess the effect of hepatic impairment relative to participants with normal hepatic function on AUC0-last an ANOVA of the log-transformed plasma PK parameters was performed. The ANOVA model included hepatic impairment as a fixed effect; Test type: Superiority or Other; p = 0.1812, ANOVA; Geometric Mean Ratio = 126.08, 95% CI 2-sided [94.59 to 168.06] — [estimate comment as in outcome 1, analysis 1]

2. Primary Outcome: Area Under the Concentration Time Curve From Time Zero Extrapolated to Infinity (AUC0-inf) of Carfilzomib 27 mg/m²
Description: The area under the curve from time zero extrapolated to infinity (AUC0-inf) following intravenous administration of carfilzomib 27 mg/m² on day 16 of cycle 1 was calculated using a non-compartmental approach, from the individual plasma concentration profiles of carfilzomib.
Time Frame: as for outcome 1
Population: Pharmacokinetic-evaluable population with data to allow terminal phase characterization
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Normal Hepatic Function | Mild Hepatic Impairment | Moderate Hepatic Impairment | Severe Hepatic Impairment
Number analyzed (Participants) | 8 | 12 | 7 | 0
ng*hr/mL | 348 (35.4) | 529 (40.3) | 500 (38.4) |
Statistical Analysis 1: Comparison: Normal Hepatic Function vs Mild Hepatic Impairment; To assess the effect of hepatic impairment relative to participants with normal hepatic function on AUC0-inf an ANOVA of the log-transformed plasma PK parameters was performed. The ANOVA model included hepatic impairment as a fixed effect; Test type: Superiority or Other; p = 0.02137, ANOVA; Geometric Mean Ratio = 151.84, 95% CI 2-sided [113.59 to 202.96] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Normal Hepatic Function vs Moderate Hepatic Impairment; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.07247, ANOVA; Geometric Mean Ratio = 143.53, 95% CI 2-sided [103.28 to 199.45] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Maximum Plasma Concentration (Cmax) of Carfilzomib 27 mg/m²
Time Frame: as for outcome 1
Population: Pharmacokinetic-evaluable population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Normal Hepatic Function | Mild Hepatic Impairment | Moderate Hepatic Impairment | Severe Hepatic Impairment
Number analyzed (Participants) | 10 | 14 | 9 | 0
ng/mL | 932 (58.4) | 1290 (47.5) | 1020 (43.7) |

4. Secondary Outcome: Time to Maximum Plasma Concentration (Tmax) of Carfilzomib 27 mg/m²
Time Frame: as for outcome 1
Population: Pharmacokinetic-evaluable population
Measure: Median (Full Range); unit: hours
Arm/Group | Normal Hepatic Function | Mild Hepatic Impairment | Moderate Hepatic Impairment | Severe Hepatic Impairment
Number analyzed (Participants) | 10 | 14 | 9 | 0
hours | 0.292 [0.250 to 0.500] | 0.458 [0.250 to 0.667] | 0.483 [0.233 to 0.750] |

5. Secondary Outcome: Clearance of Carfilzomib 27 mg/m²
Time Frame: as for outcome 1
Population: Pharmacokinetic-evaluable population with data to allow terminal phase characterization
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hour
Arm/Group | Normal Hepatic Function | Mild Hepatic Impairment | Moderate Hepatic Impairment | Severe Hepatic Impairment
Number analyzed (Participants) | 8 | 12 | 7 | 0
L/hour | 157 (32.5) | 86.4 (50.9) | 103 (43.9) |

6. Secondary Outcome: Terminal Half-life of Carfilzomib 27 mg/m²
Time Frame: as for outcome 1
Population: Pharmacokinetic-evaluable population with data to allow terminal phase characterization
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Normal Hepatic Function | Mild Hepatic Impairment | Moderate Hepatic Impairment | Severe Hepatic Impairment
Number analyzed (Participants) | 8 | 12 | 7 | 0
hours | 0.469 (22.8) | 0.541 (75.9) | 0.511 (219.4) |

7. Secondary Outcome: Mean Residence Time (MRT) of Carfilzomib 27 mg/m²
Time Frame: as for outcome 1
Population: Pharmacokinetic-evaluable population with data to allow terminal phase characterization
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Normal Hepatic Function | Mild Hepatic Impairment | Moderate Hepatic Impairment | Severe Hepatic Impairment
Number analyzed (Participants) | 8 | 12 | 7 | 0
hours | 0.108 (60.6) | 0.167 (45.7) | 0.235 (70.4) |

8. Secondary Outcome: Volume of Distribution at Steady State (Vss) of Carfilzomib 27 mg/m²
Time Frame: Cycle 1 day 16 pre-dose, 15 minutes after the start of infusion, immediately (within 2 minutes) before the end of infusion, and at 5, 15, and 30 minutes and 1, 2, and 4 hours after the end of the infusion.
Population: Pharmacokinetic-evaluable population with data to allow terminal phase characterization
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters
Arm/Group | Normal Hepatic Function | Mild Hepatic Impairment | Moderate Hepatic Impairment | Severe Hepatic Impairment
Number analyzed (Participants) | 8 | 12 | 7 | 0
liters | 16.9 (37.0) | 14.4 (58.1) | 24.2 (66.0) |

9. Secondary Outcome: Area Under the Concentration Time Curve From Time Zero to Last Concentration Measured (AUC0-last) of Carfilzomib 56 mg/m²
Description: The area under the curve from time zero to the last concentration measured (AUC0-last) following intravenous administration of carfilzomib 56 mg/m² on day 1 of cycle 2 was calculated using a non-compartmental approach, from the individual plasma concentration profiles of carfilzomib.
Time Frame: Cycle 2 day 1 pre-dose, 15 minutes after the start of infusion, immediately (within 2 minutes) before the end of infusion, and at 5, 15, and 30 minutes and 1, 2, and 4 hours after the end of the infusion.
Population: Pharmacokinetic-evaluable population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Normal Hepatic Function | Mild Hepatic Impairment | Moderate Hepatic Impairment | Severe Hepatic Impairment
Number analyzed (Participants) | 8 | 8 | 5 | 0
ng*hr/mL | 765 (100.5) | 1107 (73.7) | 927 (45.8) |

10. Secondary Outcome: Area Under the Concentration Time Curve From Time Zero Extrapolated to Infinity (AUC0-inf) of Carfilzomib 56 mg/m²
Description: The area under the curve from time zero extrapolated to infinity (AUC0-inf) following intravenous administration of carfilzomib 56 mg/m² on day 1 of cycle 2 was calculated using a non-compartmental approach, from the individual plasma concentration profiles of carfilzomib.
Time Frame: as for outcome 9
Population: Pharmacokinetic-evaluable population with data to allow terminal phase characterization
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Normal Hepatic Function | Mild Hepatic Impairment | Moderate Hepatic Impairment | Severe Hepatic Impairment
Number analyzed (Participants) | 6 | 8 | 5 | 0
ng*hr/mL | 609 (99.6) | 1108 (73.7) | 929 (46.2) |

11. Secondary Outcome: Maximum Plasma Concentration (Cmax) of Carfilzomib 56 mg/m²
Time Frame: as for outcome 9
Population: Pharmacokinetic-evaluable population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Normal Hepatic Function | Mild Hepatic Impairment | Moderate Hepatic Impairment | Severe Hepatic Impairment
Number analyzed (Participants) | 8 | 8 | 5 | 0
ng/mL | 1697 (93.7) | 2733 (67.0) | 2119 (47.9) |

12. Secondary Outcome: Time to Maximum Plasma Concentration (Tmax) of Carfilzomib 56 mg/m²
Time Frame: as for outcome 9
Population: Pharmacokinetic-evaluable population
Measure: Median (Full Range); unit: hours
Arm/Group | Normal Hepatic Function | Mild Hepatic Impairment | Moderate Hepatic Impairment | Severe Hepatic Impairment
Number analyzed (Participants) | 8 | 8 | 5 | 0
hours | 0.300 [0.250 to 0.583] | 0.408 [0.250 to 0.683] | 0.400 [0.250 to 0.583] |

13. Secondary Outcome: Terminal Half-life of Carfilzomib 56 mg/m²
Time Frame: as for outcome 9
Population: Pharmacokinetic-evaluable population with data to allow terminal phase characterization
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Normal Hepatic Function | Mild Hepatic Impairment | Moderate Hepatic Impairment | Severe Hepatic Impairment
Number analyzed (Participants) | 6 | 8 | 5 | 0
hours | 0.508 (54.7) | 0.621 (47.7) | 0.740 (137.7) |

14. Secondary Outcome: Clearance of Carfilzomib 56 mg/m²
Time Frame: as for outcome 9
Population: Pharmacokinetic-evaluable population with data to allow terminal phase characterization
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hour
Arm/Group | Normal Hepatic Function | Mild Hepatic Impairment | Moderate Hepatic Impairment | Severe Hepatic Impairment
Number analyzed (Participants) | 6 | 8 | 5 | 0
L/hour | 181 (95.9) | 92.0 (77.2) | 121 (43.5) |

15. Secondary Outcome: Mean Residence Time (MRT) of Carfilzomib 56 mg/m²
Time Frame: as for outcome 9
Population: Pharmacokinetic-evaluable population with data to allow terminal phase characterization
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Normal Hepatic Function | Mild Hepatic Impairment | Moderate Hepatic Impairment | Severe Hepatic Impairment
Number analyzed (Participants) | 6 | 8 | 5 | 0
hours | 0.0834 (195.6) | 0.161 (43.6) | 0.164 (30.7) |

16. Secondary Outcome: Volume of Distribution at Steady State (Vss) of Carfilzomib 56 mg/m²
Time Frame: as for outcome 9
Population: Pharmacokinetic-evaluable population with data to allow terminal phase characterization
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters
Arm/Group | Normal Hepatic Function | Mild Hepatic Impairment | Moderate Hepatic Impairment | Severe Hepatic Impairment
Number analyzed (Participants) | 6 | 8 | 5 | 0
liters | 15.0 (52.2) | 14.8 (51.9) | 19.8 (36.7) |

17. Secondary Outcome: Area Under the Concentration Time Curve From Time Zero to Last Concentration Measured (AUC0-last) for Metabolite PR-389/M14
Time Frame: Cycle 1 day 16 and cycle 2 day 1 pre-dose, 15 minutes after the start of infusion, immediately (within 2 minutes) before the end of infusion, and at 5, 15, and 30 minutes and 1, 2, and 4 hours after the end of the infusion.
Population: Pharmacokinetic-evaluable population, defined as all participants who had adequate carfilzomib exposure and plasma concentration versus time data for the estimation of PK parameters by a non-compartmental analysis at each time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Normal Hepatic Function | Mild Hepatic Impairment | Moderate Hepatic Impairment | Severe Hepatic Impairment
Number analyzed (Participants) | 10 | 14 | 9 | 0
ng*hr/mL
  Cycle 1 Day 16 (27 mg/m²); N = 10, 14, 9, 0 | 463 (42.5) | 417 (30.5) | 385 (26.8) |
  Cycle 2 Day 1 (56 mg/m²); N = 8, 8, 5, 0 | 837 (26.8) | 752 (29.7) | 786 (20.3) |

18. Secondary Outcome: Area Under the Concentration Time Curve From Time Zero Extrapolated to Infinity (AUC0-inf) for Metabolite PR-389/M14
Time Frame: as for outcome 17
Population: Pharmacokinetic-evaluable population with data to allow terminal phase characterization
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Normal Hepatic Function | Mild Hepatic Impairment | Moderate Hepatic Impairment | Severe Hepatic Impairment
Number analyzed (Participants) | 4 | 11 | 8 | 0
ng*hr/mL
  Cycle 1 Day 16 (27 mg/m²); N = 4, 11, 8, 0 | 400 (19.3) | 432 (29.9) | 437 (32.7) |
  Cycle 2 Day 1 (56 mg/m²); N = 4, 6, 5, 0 | 834 (6.3) | 770 (27.2) | 843 (22.3) |

19. Secondary Outcome: Maximum Plasma Concentration (Cmax) for Metabolite PR-389/M14
Time Frame: as for outcome 17
Population: Pharmacokinetic-evaluable population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Normal Hepatic Function | Mild Hepatic Impairment | Moderate Hepatic Impairment | Severe Hepatic Impairment
Number analyzed (Participants) | 10 | 14 | 9 | 0
ng/mL
  Cycle 1 Day 16 (27 mg/m²); N = 10, 14, 9, 0 | 189 (32.5) | 198 (22.7) | 201 (26.5) |
  Cycle 2 Day 1 (56 mg/m²); N = 8, 8, 5, 0 | 381 (15.0) | 345 (25.9) | 513 (24.3) |

20. Secondary Outcome: Time to Maximum Plasma Concentration (Tmax) for Metabolite PR-389/M14
Time Frame: as for outcome 17
Population: Pharmacokinetic-evaluable population
Measure: Median (Full Range); unit: hours
Arm/Group | Normal Hepatic Function | Mild Hepatic Impairment | Moderate Hepatic Impairment | Severe Hepatic Impairment
Number analyzed (Participants) | 10 | 14 | 9 | 0
hours
  Cycle 1 Day 16 (27 mg/m²); N = 10, 14, 9, 0 | 0.867 [0.583 to 1.52] | 0.792 [0.633 to 1.50] | 0.750 [0.583 to 1.00] |
  Cycle 2 Day 1 (56 mg/m²); N = 8, 8, 5, 0 | 0.842 [0.750 to 1.48] | 0.992 [0.750 to 1.60] | 0.750 [0.650 to 0.783] |

21. Secondary Outcome: Terminal Half-life for Metabolite PR-389/M14
Time Frame: as for outcome 17
Population: Pharmacokinetic-evaluable population with data to allow terminal phase characterization
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Normal Hepatic Function | Mild Hepatic Impairment | Moderate Hepatic Impairment | Severe Hepatic Impairment
Number analyzed (Participants) | 4 | 11 | 8 | 0
hours
  Cycle 1 Day 16 (27 mg/m²); N = 4, 11, 8, 0 | 1.42 (10.3) | 1.20 (13.7) | 1.26 (18.0) |
  Cycle 2 Day 1 (56 mg/m²); N = 4, 6, 5, 0 | 1.32 (15.3) | 1.30 (16.1) | 1.07 (13.6) |

22. Secondary Outcome: Mean Residence Time (MRT) for Metabolite PR-389/M14
Time Frame: as for outcome 17
Population: Pharmacokinetic-evaluable population with data to allow terminal phase characterization
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Normal Hepatic Function | Mild Hepatic Impairment | Moderate Hepatic Impairment | Severe Hepatic Impairment
Number analyzed (Participants) | 4 | 11 | 8 | 0
hours
  Cycle 1 Day 16 (27 mg/m²); N = 4, 11, 8, 0 | 2.42 (11.4) | 2.13 (12.2) | 2.14 (16.0) |
  Cycle 2 Day 1 (56 mg/m²); N = 4, 6, 5, 0 | 2.25 (10.8) | 2.27 (15.8) | 1.78 (11.2) |

23. Secondary Outcome: Area Under the Concentration Time Curve From Time Zero to Last Concentration Measured (AUC0-last) for Metabolite PR-413/M15
Time Frame: as for outcome 17
Population: Pharmacokinetic-evaluable population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Normal Hepatic Function | Mild Hepatic Impairment | Moderate Hepatic Impairment | Severe Hepatic Impairment
Number analyzed (Participants) | 10 | 14 | 9 | 0
ng*hr/mL
  Cycle 1 Day 16 (27 mg/m²); N = 10, 14, 9, 0 | 50.1 (39.5) | 56.7 (33.9) | 85.5 (36.6) |
  Cycle 2 Day 1 (56 mg/m²); N = 8, 8, 5, 0 | 106 (33.7) | 119 (38.9) | 173 (17.8) |

24. Secondary Outcome: Area Under the Concentration Time Curve From Time Zero Extrapolated to Infinity (AUC0-inf) for Metabolite PR-413/M15
Time Frame: as for outcome 17
Population: Pharmacokinetic-evaluable population with data to allow terminal phase characterization
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Normal Hepatic Function | Mild Hepatic Impairment | Moderate Hepatic Impairment | Severe Hepatic Impairment
Number analyzed (Participants) | 10 | 13 | 8 | 0
ng*hr/mL
  Cycle 1 Day 16 (27 mg/m²); N = 10, 13, 8, 0 | 56.6 (43.7) | 60.8 (32.6) | 92.9 (41.7) |
  Cycle 2 Day 1 (56 mg/m²); N = 8, 8, 5, 0 | 116 (36.9) | 132 (41.0) | 186 (18.2) |

25. Secondary Outcome: Maximum Plasma Concentration (Cmax) for Metabolite PR-413/M15
Time Frame: as for outcome 17
Population: Pharmacokinetic-evaluable population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Normal Hepatic Function | Mild Hepatic Impairment | Moderate Hepatic Impairment | Severe Hepatic Impairment
Number analyzed (Participants) | 10 | 14 | 9 | 0
ng/mL
  Cycle 1 Day 16 (27 mg/m²); N = 10, 14, 9, 0 | 27.8 (30.5) | 33.9 (30.7) | 46.3 (26.6) |
  Cycle 2 Day 1 (56 mg/m²); N = 8, 8, 5, 0 | 59.4 (27.5) | 66.0 (37.2) | 103 (19.5) |

26. Secondary Outcome: Time to Maximum Plasma Concentration (Tmax) for Metabolite PR-413/M15
Time Frame: as for outcome 17
Population: Pharmacokinetic-evaluable population
Measure: Median (Full Range); unit: hours
Arm/Group | Normal Hepatic Function | Mild Hepatic Impairment | Moderate Hepatic Impairment | Severe Hepatic Impairment
Number analyzed (Participants) | 10 | 14 | 9 | 0
hours
  Cycle 1 Day 16 (27 mg/m²); N = 10, 14, 9, 0 | 0.750 [0.583 to 0.767] | 0.767 [0.583 to 1.00] | 0.650 [0.583 to 1.10] |
  Cycle 2 Day 1 (56 mg/m²); N = 8, 8, 5, 0 | 0.717 [0.600 to 1.00] | 0.800 [0.467 to 1.08] | 0.750 [0.617 to 0.750] |

27. Secondary Outcome: Terminal Half-life for Metabolite PR-413/M15
Time Frame: as for outcome 17
Population: Pharmacokinetic-evaluable population with data to allow terminal phase characterization
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Normal Hepatic Function | Mild Hepatic Impairment | Moderate Hepatic Impairment | Severe Hepatic Impairment
Number analyzed (Participants) | 10 | 13 | 8 | 0
hours
  Cycle 1 Day 16 (27 mg/m²); N = 10, 13, 8, 0 | 1.34 (18.9) | 1.25 (13.6) | 1.23 (17.6) |
  Cycle 2 Day 1 (56 mg/m²); N = 8, 8, 5, 0 | 1.18 (21.8) | 1.24 (10.2) | 1.07 (16.0) |

28. Secondary Outcome: Mean Residence Time (MRT) for Metabolite PR-413/M15
Time Frame: as for outcome 17
Population: Pharmacokinetic-evaluable population with data to allow terminal phase characterization
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Normal Hepatic Function | Mild Hepatic Impairment | Moderate Hepatic Impairment | Severe Hepatic Impairment
Number analyzed (Participants) | 10 | 13 | 8 | 0
hours
  Cycle 1 Day 16 (27 mg/m²); N = 10, 13, 8, 0 | 2.13 (15.8) | 2.02 (8.8) | 2.04 (14.6) |
  Cycle 2 Day 1 (56 mg/m²); N = 8, 8, 5, 0 | 1.96 (18.9) | 2.09 (8.0) | 1.83 (8.9) |

29. Secondary Outcome: Area Under the Concentration Time Curve From Time Zero to Last Concentration Measured (AUC0-last) for Metabolite PR-519/M16
Time Frame: as for outcome 17
Population: Pharmacokinetic-evaluable population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Normal Hepatic Function | Mild Hepatic Impairment | Moderate Hepatic Impairment | Severe Hepatic Impairment
Number analyzed (Participants) | 10 | 14 | 9 | 0
ng*hr/mL
  Cycle 1 Day 16 (27 mg/m²); N = 10, 14, 9, 0 | 125 (27.6) | 136 (45.2) | 228 (37.3) |
  Cycle 2 Day 1 (56 mg/m²); N = 8, 8, 5, 0 | 278 (23.4) | 311 (42.9) | 463 (24.5) |

30. Secondary Outcome: Area Under the Concentration Time Curve From Time Zero Extrapolated to Infinity (AUC0-inf) for Metabolite PR-519/M16
Time Frame: as for outcome 17
Population: Pharmacokinetic-evaluable population with data to allow terminal phase characterization
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Normal Hepatic Function | Mild Hepatic Impairment | Moderate Hepatic Impairment | Severe Hepatic Impairment
Number analyzed (Participants) | 10 | 14 | 8 | 0
ng*hr/mL
  Cycle 1 Day 16 (27 mg/m²); N = 10, 14, 8, 0 | 127 (27.8) | 138 (44.9) | 235 (39.4) |
  Cycle 2 Day 1 (56 mg/m²); N = 7, 8, 5, 0 | 281 (25.6) | 314 (42.7) | 465 (24.4) |

31. Secondary Outcome: Maximum Plasma Concentration (Cmax) for Metabolite PR-519/M16
Time Frame: as for outcome 17
Population: Pharmacokinetic-evaluable population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Normal Hepatic Function | Mild Hepatic Impairment | Moderate Hepatic Impairment | Severe Hepatic Impairment
Number analyzed (Participants) | 10 | 14 | 9 | 0
ng/mL
  Cycle 1 Day 16 (27 mg/m²); N = 10, 14, 9, 0 | 145 (30.7) | 160 (42.0) | 257 (43.6) |
  Cycle 2 Day 1 (56 mg/m²); N = 8, 8, 5, 0 | 314 (33.6) | 349 (39.5) | 546 (23.4) |

32. Secondary Outcome: Time to Maximum Plasma Concentration (Tmax) for Metabolite PR-519/M16
Time Frame: as for outcome 17
Population: Pharmacokinetic-evaluable population
Measure: Median (Full Range); unit: hours
Arm/Group | Normal Hepatic Function | Mild Hepatic Impairment | Moderate Hepatic Impairment | Severe Hepatic Impairment
Number analyzed (Participants) | 10 | 14 | 9 | 0
hours
  Cycle 1 Day 16 (27 mg/m²); N = 10, 14, 9, 0 | 0.500 [0.250 to 0.667] | 0.600 [0.250 to 0.750] | 0.700 [0.583 to 0.850] |
  Cycle 2 Day 1 (56 mg/m²); N = 8, 8, 5, 0 | 0.483 [0.250 to 0.617] | 0.592 [0.250 to 0.850] | 0.583 [0.467 to 0.650] |

33. Secondary Outcome: Terminal Half-life for Metabolite PR-519/M16
Time Frame: as for outcome 17
Population: Pharmacokinetic-evaluable population with data to allow terminal phase characterization
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Normal Hepatic Function | Mild Hepatic Impairment | Moderate Hepatic Impairment | Severe Hepatic Impairment
Number analyzed (Participants) | 10 | 14 | 8 | 0
hours
  Cycle 1 Day 16 (27 mg/m²); N = 10, 14, 8, 0 | 0.786 (14.0) | 0.728 (22.6) | 0.673 (13.6) |
  Cycle 2 Day 1 (56 mg/m²); N = 7, 8, 5, 0 | 0.748 (22.2) | 0.680 (10.7) | 0.601 (8.2) |

34. Secondary Outcome: Mean Residence Time (MRT) for Metabolite PR-519/M16
Time Frame: as for outcome 17
Population: Pharmacokinetic-evaluable population with data to allow terminal phase characterization
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Normal Hepatic Function | Mild Hepatic Impairment | Moderate Hepatic Impairment | Severe Hepatic Impairment
Number analyzed (Participants) | 10 | 14 | 8 | 0
hours
  Cycle 1 Day 16 (27 mg/m²); N = 10, 14, 8, 0 | 1.01 (11.3) | 0.961 (29.1) | 0.994 (13.3) |
  Cycle 2 Day 1 (56 mg/m²); N = 8, 8, 5, 0 | 0.994 (9.0) | 1.00 (14.2) | 0.909 (7.8) |

35. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: Treatment-related adverse events (TRAEs) are adverse events considered related to carfilzomib by the investigator, including those with unknown relationship.
  Adverse events were graded using National Cancer Institute's Common Terminology Criteria for Adverse Events (NCI-CTCAE), version 4.03, on a scale from 1 (mild) to 5 (death).
Time Frame: From the first dose of carfilzomib until 30 days after last dose; the overall median duration of treatment was 4.2 weeks
Measure: Number; unit: participants
Arm/Group | Normal Hepatic Function | Mild Hepatic Impairment | Moderate Hepatic Impairment | Severe Hepatic Impairment
Number analyzed (Participants) | 11 | 17 | 14 | 4
participants
  Any adverse event | 10 | 17 | 14 | 4
  Adverse event Grade ≥ 3 | 7 | 12 | 13 | 3
  Serious adverse events | 3 | 10 | 8 | 4
  Leading to discontinuation of carfilzomib | 1 | 2 | 4 | 0
  Fatal adverse events | 1 | 4 | 1 | 3
  Treatment-related adverse events (TRAE) | 8 | 13 | 12 | 1
  Treatment-related adverse events Grade ≥ 3 | 2 | 5 | 8 | 0
  Treatment-related serious adverse events | 0 | 3 | 4 | 0
  TRAE leading to discontinuation of carfilzomib | 1 | 0 | 3 | 0
  Treatment-related fatal adverse events | 0 | 2 | 0 | 0

ADVERSE EVENTS:
Time Frame: From the first dose of carfilzomib until 30 days after last dose; the overall median duration of treatment was 4.2 weeks.
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Arm/Group | Normal Hepatic Function | Mild Hepatic Impairment | Moderate Hepatic Impairment | Severe Hepatic Impairment
Serious Adverse Events (participants affected / at risk) | 3/11 | 10/17 | 8/14 | 4/4
Other Adverse Events (participants affected / at risk) | 10/11 | 17/17 | 14/14 | 3/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Normal Hepatic Function (N=11) | Mild Hepatic Impairment (N=17) | Moderate Hepatic Impairment (N=14) | Severe Hepatic Impairment (N=4)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0
Splenic vein occlusion (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 3 | 0
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastric varices haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Oral cavity fistula (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Disease progression (General disorders) | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 0
Multi-organ failure (General disorders) | 0 | 0 | 0 | 1
Acute hepatic failure (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Bacterial sepsis (Infections and infestations) | 0 | 0 | 0 | 1
Biliary sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 1 | 0 | 0
Sepsis (Infections and infestations) | 1 | 1 | 1 | 0
Septic shock (Infections and infestations) | 0 | 0 | 0 | 1
Viral infection (Infections and infestations) | 0 | 1 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 2 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hepatic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 2
Spinal cord compression (Nervous system disorders) | 1 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1 | 2
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Normal Hepatic Function (N=11) | Mild Hepatic Impairment (N=17) | Moderate Hepatic Impairment (N=14) | Severe Hepatic Impairment (N=4)
Anaemia (Blood and lymphatic system disorders) | 6 | 10 | 3 | 2
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 4 | 0
Left ventricular dysfunction (Cardiac disorders) | 1 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Eye discharge (Eye disorders) | 1 | 0 | 0 | 0
Lacrimation increased (Eye disorders) | 1 | 0 | 0 | 0
Ocular icterus (Eye disorders) | 0 | 0 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 1 | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 3 | 4 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 1 | 1 | 1
Constipation (Gastrointestinal disorders) | 1 | 5 | 4 | 0
Diarrhoea (Gastrointestinal disorders) | 4 | 4 | 4 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Epigastric discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Faecal incontinence (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 2 | 0 | 0
Hyperchlorhydria (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Melaena (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 3 | 5 | 5 | 0
Retching (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 3 | 2 | 3 | 0
Asthenia (General disorders) | 1 | 0 | 1 | 0
Chest pain (General disorders) | 1 | 0 | 0 | 0
Chills (General disorders) | 2 | 0 | 2 | 0
Early satiety (General disorders) | 0 | 1 | 0 | 0
Face oedema (General disorders) | 0 | 1 | 0 | 0
Fatigue (General disorders) | 8 | 7 | 8 | 0
General physical health deterioration (General disorders) | 0 | 0 | 1 | 0
Infusion site discomfort (General disorders) | 0 | 1 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0 | 0
Oedema peripheral (General disorders) | 4 | 2 | 5 | 0
Pyrexia (General disorders) | 1 | 1 | 2 | 0
Temperature intolerance (General disorders) | 1 | 0 | 0 | 0
Thirst (General disorders) | 0 | 1 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 3 | 2 | 0
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0
Candida infection (Infections and infestations) | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 1 | 0
Liver abscess (Infections and infestations) | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 1 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 5 | 4 | 0
Ammonia increased (Investigations) | 0 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 4 | 4 | 0
Basophil count increased (Investigations) | 1 | 0 | 0 | 0
Blood albumin decreased (Investigations) | 1 | 0 | 0 | 0
Blood alkaline phosphatase decreased (Investigations) | 0 | 1 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 1 | 2 | 0
Blood bicarbonate decreased (Investigations) | 0 | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 1 | 9 | 0
Blood calcium decreased (Investigations) | 0 | 1 | 0 | 0
Blood creatinine increased (Investigations) | 2 | 1 | 1 | 0
Blood lactate dehydrogenase increased (Investigations) | 1 | 1 | 1 | 0
Blood potassium increased (Investigations) | 1 | 0 | 0 | 0
Blood urea increased (Investigations) | 1 | 0 | 1 | 0
Creatinine renal clearance decreased (Investigations) | 0 | 1 | 0 | 0
Haematocrit decreased (Investigations) | 1 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 2 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 1 | 0 | 0
Monocyte count increased (Investigations) | 1 | 0 | 0 | 0
Platelet count decreased (Investigations) | 1 | 1 | 0 | 0
Red blood cell count decreased (Investigations) | 1 | 0 | 0 | 0
Urine output decreased (Investigations) | 0 | 0 | 1 | 0
Weight decreased (Investigations) | 2 | 2 | 0 | 0
White blood cell count increased (Investigations) | 1 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 3 | 5 | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 | 3 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 2 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 2 | 1 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 2 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0
Malnutrition (Metabolism and nutrition disorders) | 1 | 1 | 1 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 2 | 1 | 3 | 0
Dizziness postural (Nervous system disorders) | 1 | 0 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 3 | 1 | 2 | 0
Lethargy (Nervous system disorders) | 1 | 3 | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 1 | 1 | 0 | 0
Restless legs syndrome (Nervous system disorders) | 1 | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 1 | 1 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 3 | 1 | 2 | 0
Mental disorder (Psychiatric disorders) | 1 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0 | 0
Cystitis noninfective (Renal and urinary disorders) | 0 | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 1 | 0 | 0
Renal pain (Renal and urinary disorders) | 0 | 0 | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 4 | 3 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 2 | 2 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Skin oedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 2 | 0 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 1 | 1
Orthostatic hypotension (Vascular disorders) | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.